CLINICAL TRIAL: NCT02714335
Title: An Observational Study to Determine the Correlation Between MAGE-A3, PRAME Polymorphism and Expression Levels of MAGE-A3 and PRAME in NSCLC Patients in Taiwan
Brief Title: The Correlation Between MAGE-A3, PRAME Polymorphism and Expression Levels of MAGE-A3 and PRAME in NSCLC Patients
Status: Completed | Type: Observational
Sponsor: Szu-Hua Pan (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Szu-Hua Pan, Dr., National Taiwan University
Organization: National Taiwan University (Other)
Other Study IDs: 114764
Record Dates: First submitted 2016-03-02; First posted 2016-03-21 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Considering the low expression rate of Melanoma-associated antigen 3 (MAGE-A3) in Asian especially Southeast Asian, it would be great interests to investigate the potential polymorphism of MAGE-A3 in Non-Small-Cell Lung Cancer (NSCLC) patients in Taiwan. Meanwhile, it is also interesting to study the expression of Preferentially Expressed Antigen In Melanoma(PRAME) and Epidermal growth factor receptor (EGFR) mutation status as well as to find out significant factors which may affect their expression such as smoking status, histological types, tumour size and stages in Taiwan.

DETAILED DESCRIPTION:
Considering the low expression rate of MAGE-A3 in Asian especially Southeast Asian, it would be great interests to investigate the potential polymorphism of MAGE-A3 in NSCLC patients in Taiwan. Meanwhile, it is also interesting to study the expression of PRAME and EGFR mutation status as well as to find out significant factors which may affect their expression such as smoking status, histological types, tumour size and stages in Taiwan

ELIGIBILITY:
Inclusion Criteria:

- Tissues samples up to 200 cases of NSCLS patients with informed consent, consisting of about 100 cases of adenocarcinoma (AC) and 100 cases of squamous cell carcinoma (SCC), with stage of IB, IIA, IIB and IIIA

Exclusion Criteria:

- No

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Site will retrieve tissue samples of around 200 cases of NSCLC patients with informed consent including about 100 cases of adenocarcinoma (AC) and 100 cases of squamous cell carcinoma (SCC), with stages of IB, IIA, IIB and IIIA.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least one MAGE-A3 gene single nucleotide polymorphism (SNP) | up to 44 months

IPD SHARING:
Plan to Share IPD: Yes
• Type of publication e.g. poster, abstract, oral presentation etc. Poster and original article